CLINICAL TRIAL: NCT01765777
Title: Efficacy of Osteopathic Manipulative Medicine (OMM) and Phototherapy for Patients With Chronic Lower Back Pain
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: New York Institute of Technology (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: BHS-740
Record Dates: First submitted 2013-01-08; First posted 2013-01-10 (Estimated); Last update posted 2024-08-06 (Actual); Status verified 2024-08

CONDITIONS: Chronic Lower Back Pain
Keywords: Low back pain; Lower back pain; Chronic back pain
MeSH Terms: conditions — Low Back Pain | interventions — Phototherapy; Low-Level Light Therapy

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- Control Group (No Intervention): Subjects in this arm continue with standard medical care
- Osteopathic Manipulative Medicine Group (Experimental): Subjects in this arm will receive an OMM intervention.
  Interventions: Procedure: Osteopathic Manipulative Medicine
- Phototherapy Group (Experimental): Subjects in this arm will receive a phototherapy intervention.
  Interventions: Procedure: Phototherapy
- OMM and Phototherapy Group (Experimental): Subjects in this arm will receive both the OMM and phototherapy interventions.
  Interventions: Procedure: Osteopathic Manipulative Medicine; Procedure: Phototherapy

INTERVENTIONS:
Procedure: Osteopathic Manipulative Medicine
  Other Names: OMM,OMT
  Arms: OMM and Phototherapy Group; Osteopathic Manipulative Medicine Group
Procedure: Phototherapy
  Other Names: Low level laser therapy; LLLT
  Arms: OMM and Phototherapy Group; Phototherapy Group

SUMMARY:
The purpose of the research study entitled "Efficacy of Osteopathic Manipulative Medicine (OMM) and Phototherapy for Patients with Chronic Lower Back Pain" is to investigate the hypothesis that combined treatment with both osteopathic manipulative medicine (OMM) and phototherapy will provide greater pain relief for patients with chronic lower back pain, as compared with standard medical management or either treatment alone.

DETAILED DESCRIPTION:
The research has demonstrated separately that phototherapy and osteopathic manipulative medicine (OMM) are effective in reducing chronic low back pain, However there has not been any research to evaluate whether the interaction of the two treatment approaches together can provide enhanced pain relief. In A Meta-analysis of the Efficacy of Phototherapy in Tissue Repair, Fulop et.al.(1) from the Department of Physical Therapy, School of Health Professions, New York Institute of Technology (NYIT) concluded that "phototherapy is a highly effective form of treatment for tissue repair, with stronger supporting evidence resulting from experimental animal studies than human studies" (Fulop, p. 695, 699). Further review of the literature by Fulop et. al. (2) focused on the question of pain relief in relation to phototherapy, and the conclusion was that pain from various etiologies can be effectively relieved by phototherapy. The U.S. Food and Drug Administration has cleared biostimulation lasers (a.k.a. low level laser therapy [LLLT], cold lasers, soft lasers, or laser acupuncture devices) for marketing as "adjunctive devices for the temporary relief of pain" (3). Thus, both health practitioners and the lay public have access to and may potentially obtain and use phototherapy devices manufactured by various companies. Other research protocols by Gur, A et. al. (4) and Djavid, GE et. al. (5) evaluated patients with chronic low back pain in relation to the combined effectiveness of low level laser therapy and exercise. These studies showed positive results with the combined approaches.

Osteopathic physicians utilize an approach to the treatment of patients called osteopathic manipulative medicine (OMM). The osteopathic physician will diagnose somatic dysfunction, and then treat the dysfunctions found with one or more of several OMM treatment approaches. The American Osteopathic Association (AOA) published in 2009 the "Guidelines for Osteopathic Manipulative Treatment (OMT) for Patients with Low Back Pain." These guidelines are available both through the AOA and the Agency for Healthcare Research and Quality (AHRQ), National Guideline Clearinghouse (6). This guideline (6) specifically addresses the "efficacy of osteopathic manipulation treatment in reducing low back pain" (p. 2). A review of the literature was performed, and after selection a total of "six trials, involving eight osteopathic manipulative treatment (OMT) vs control treatment comparisons, were included" in the meta-analysis (p. 2-3). The major recommendation stated in the guideline is that "osteopathic manipulative treatment (OMT) be utilized by osteopathic physicians for musculoskeletal causes of back pain, i.e., to treat the diagnoses of somatic dysfunctions related to the low back pain" (p.4). In addition, the meta-analysis performed did show that OMT for patients with low back pain led to statistically significant reduction in pain (p. 5). Thus, the potential for a complementary approach to patient care in cases of chronic low back pain exists. Yet, no studies to date have specifically evaluated this particular hypothesis regarding OMT and phototherapy for patients with chronic low back pain. The purpose of this research is to evaluate this question of enhanced combined efficacy for the overall benefit of patients.

ELIGIBILITY:
Inclusion Criteria:

* Age range: 18 - 65 years old
* Subjects with constant or intermittent nonspecific lower back pain for a minimum of three (3) months duration.

Exclusion Criteria:

* Prospective subjects with a diagnosis of the following potential underlying causes of lower back pain: ankylosing spondylitis, cancer or a history of a histologically demonstrated malignant carcinoma, cauda equine syndrome, herniated disc, spinal fracture, or spinal osteomyelitis.
* Prospective subjects who have undergone surgery of the lower back in the preceding three (3) months.
* Prospective subjects who have received worker's compensation in the preceding three (3) months, or are involved in litigation involving concerns of lower back.
* Prospective subjects who are pregnant.
* Prospective subjects who have been a patient receiving any osteopathic manipulative medicine (OMM) treatment at the clinical trial site in the previous three (3) months, or on greater than three (3) occasions in the preceding year.
* Prospective subjects who have ever been an employee at the clinical trial site.
* Prospective subjects who have received spinal manipulation in the previous three (3) months, or on greater than three (3) occasions in the preceding year.
* Prospective subjects who are currently involved in a physical therapy rehabilitation program.
* Prospective subjects who have photosensitivity.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2011-06 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
10 cm visual analog scale for quantitative back pain | 8 weeks
  VAS Data collected at all visits
SF-36 Health Survey to measure Quality of Life | 8 weeks
  SF-36 survey data collected at 3 points
The Oswestry Back Questionnaire to measure qualitative back pain | 8 weeks
  Oswestry questionnaire data collected at 3 points

CONTACTS AND LOCATIONS:
Overall Officials: Patricia S Kooyman, D.O., Principal Investigator — New York Institute of Technology
Locations (1):
- New York Institute of Technology, Old Westbury, New York, United States

REFERENCES:
- [Background] Fulop AM, Dhimmer S, Deluca JR, Johanson DD, Lenz RV, Patel KB, Douris PC, Enwemeka CS. A meta-analysis of the efficacy of phototherapy in tissue repair. Photomed Laser Surg. 2009 Oct;27(5):695-702. doi: 10.1089/pho.2009.2550. PMID 19698019
- [Background] Gur A, Karakoc M, Cevik R, Nas K, Sarac AJ, Karakoc M. Efficacy of low power laser therapy and exercise on pain and functions in chronic low back pain. Lasers Surg Med. 2003;32(3):233-8. doi: 10.1002/lsm.10134. PMID 12605431
- [Background] Djavid GE, Mehrdad R, Ghasemi M, Hasan-Zadeh H, Sotoodeh-Manesh A, Pouryaghoub G. In chronic low back pain, low level laser therapy combined with exercise is more beneficial than exercise alone in the long term: a randomised trial. Aust J Physiother. 2007;53(3):155-60. doi: 10.1016/s0004-9514(07)70022-3. PMID 17725472
- [Background] Licciardone JC, Stoll ST, Fulda KG, Russo DP, Siu J, Winn W, Swift J Jr. Osteopathic manipulative treatment for chronic low back pain: a randomized controlled trial. Spine (Phila Pa 1976). 2003 Jul 1;28(13):1355-62. doi: 10.1097/01.BRS.0000067110.61471.7D. PMID 12838090
- [Background] Williams NH, Wilkinson C, Russell I, Edwards RT, Hibbs R, Linck P, Muntz R. Randomized osteopathic manipulation study (ROMANS): pragmatic trial for spinal pain in primary care. Fam Pract. 2003 Dec;20(6):662-9. doi: 10.1093/fampra/cmg607. PMID 14701889
- [Background] Williams N. Managing back pain in general practice--is osteopathy the new paradigm? Br J Gen Pract. 1997 Oct;47(423):653-5. PMID 9474832
- [Background] Ferreira ML, Ferreira PH, Latimer J, Herbert RD, Hodges PW, Jennings MD, Maher CG, Refshauge KM. Comparison of general exercise, motor control exercise and spinal manipulative therapy for chronic low back pain: A randomized trial. Pain. 2007 Sep;131(1-2):31-7. doi: 10.1016/j.pain.2006.12.008. Epub 2007 Jan 23. PMID 17250965
- [Background] Burton AK, McClune TD, Clarke RD, Main CJ. Long-term follow-up of patients with low back pain attending for manipulative care: outcomes and predictors. Man Ther. 2004 Feb;9(1):30-5. doi: 10.1016/s1356-689x(03)00052-3. PMID 14723859
- [Background] Harvey E, Burton AK, Moffett JK, Breen A; UK BEAM trial team. Spinal manipulation for low-back pain: a treatment package agreed to by the UK chiropractic, osteopathy and physiotherapy professional associations. Man Ther. 2003 Feb;8(1):46-51. doi: 10.1054/math.2002.0472. PMID 12635637
- [Background] Kimberly PE. Formulating a prescription for osteopathic manipulative treatment. J Am Osteopath Assoc. 1980 Apr;79(8):506-13. No abstract available. PMID 7364595
- [Background] Ramirez MA, Haman J, Worth L. Low back pain: diagnosis by six newly discovered sacral tender points and treatment with counterstrain. J Am Osteopath Assoc. 1989 Jul;89(7):905-6, 911-3. PMID 2527838
- [Background] Hoffman KS, Hoffman LL. Effects of adding sacral base leveling to osteopathic manipulative treatment of back pain: a pilot study. J Am Osteopath Assoc. 1994 Mar;94(3):217-20, 223-6. PMID 8200825
- [Background] Jokl P. Twenty-eighth annual AOA/NOF Research Conference, 1984: part I. Keynote address: Muscle and low-back pain. J Am Osteopath Assoc. 1984 Sep;84(1):64-6. No abstract available. PMID 6238015
- [Background] Hoyt WH, Bard DA, Shaffer F. Experience with an antigravity leverage device for chronic low back pain: a clinical study. J Am Osteopath Assoc. 1981 Mar;80(7):474-9. No abstract available. PMID 6453859
- [Background] Korr IM. The spinal cord as organizer of disease processes: IV. Axonal transport and neurotrophic function in relation to somatic dysfunction. J Am Osteopath Assoc. 1981 Mar;80(7):451-9. No abstract available. PMID 6263830
- [Background] Licciardone JC. The unique role of osteopathic physicians in treating patients with low back pain. J Am Osteopath Assoc. 2004 Nov;104(11 Suppl 8):S13-8. PMID 15602036
- [Background] Nadler SF. Nonpharmacologic management of pain. J Am Osteopath Assoc. 2004 Nov;104(11 Suppl 8):S6-12. PMID 15602035
- [Background] Hoehler FK, Tobis JS, Buerger AA. Spinal manipulation for low back pain. JAMA. 1981 May 8;245(18):1835-8. PMID 6453240
- [Background] Niemisto L, Sarna S, Lahtinen-Suopanki T, Lindgren KA, Hurri H. Predictive factors for 1-year outcome of chronic low back pain following manipulation, stabilizing exercises, and physician consultation or physician consultation alone. J Rehabil Med. 2004 May;36(3):104-9. doi: 10.1080/16501970310019151. PMID 15209452
- [Background] Tong HC, Heyman OG, Lado DA, Isser MM. Interexaminer reliability of three methods of combining test results to determine side of sacral restriction, sacral base position, and innominate bone position. J Am Osteopath Assoc. 2006 Aug;106(8):464-8. PMID 16943516
- [Background] Snider KT, Johnson JC, Snider EJ, Degenhardt BF. Increased incidence and severity of somatic dysfunction in subjects with chronic low back pain. J Am Osteopath Assoc. 2008 Aug;108(8):372-8. PMID 18723455
- [Background] Andersson GB, Lucente T, Davis AM, Kappler RE, Lipton JA, Leurgans S. A comparison of osteopathic spinal manipulation with standard care for patients with low back pain. N Engl J Med. 1999 Nov 4;341(19):1426-31. doi: 10.1056/NEJM199911043411903. PMID 10547405
- [Background] Gamber R, Holland S, Russo DP, Cruser dA, Hilsenrath PE. Cost-effective osteopathic manipulative medicine: a literature review of cost-effectiveness analyses for osteopathic manipulative treatment. J Am Osteopath Assoc. 2005 Aug;105(8):357-67. PMID 16166390
- [Background] McPartland JM, Giuffrida A, King J, Skinner E, Scotter J, Musty RE. Cannabimimetic effects of osteopathic manipulative treatment. J Am Osteopath Assoc. 2005 Jun;105(6):283-91. PMID 16118355
- [Background] Licciardone JC, Russo DP. Blinding protocols, treatment credibility, and expectancy: methodologic issues in clinical trials of osteopathic manipulative treatment. J Am Osteopath Assoc. 2006 Aug;106(8):457-63. PMID 16943515
- [Background] Wearn AM, Greenfield SM. Access to complementary medicine in general practice: survey in one UK health authority. J R Soc Med. 1998 Sep;91(9):465-70. doi: 10.1177/014107689809100904. PMID 9849516
- [Background] Mein EA, Greenman PE, McMillin DL, Richards DG, Nelson CD. Manual medicine diversity: research pitfalls and the emerging medical paradigm. J Am Osteopath Assoc. 2001 Aug;101(8):441-4. PMID 11526876
- [Background] Navratil L, Kymplova J. Contraindications in noninvasive laser therapy: truth and fiction. J Clin Laser Med Surg. 2002 Dec;20(6):341-3. doi: 10.1089/104454702320901134. PMID 12513921
- [Background] Fulop AM, Dhimmer S, Deluca JR, Johanson DD, Lenz RV, Patel KB, Douris PC, Enwemeka CS. A meta-analysis of the efficacy of laser phototherapy on pain relief. Clin J Pain. 2010 Oct;26(8):729-36. doi: 10.1097/AJP.0b013e3181f09713. PMID 20842007
- [Background] Patterson, MM, PhD, Editorial - Research in OMT: What is the question and do we understand it?, JAOA, January 2007, Vol. 107, No. 1, pp. 8-11.
- [Background] Cameron, Michelle H., Physical Agents in Rehabilitation: From Research to Practice, Third Edition, Chapter 12, Electromagnetic Radiation: Lasers and Light, Saunders Elsevier, 2009.
- [Background] Task Force on the Low Back Pain Clinical Practice Guidelines. American Osteopathic Association Guidelines for Osteopathic Manipulative Treatment (OMT) for Patients With Low Back Pain. J Am Osteopath Assoc. 2016 Aug 1;116(8):536-49. doi: 10.7556/jaoa.2016.107. PMID 27455103
- See also: AHRQ - American Osteopathic Association guidelines for osteopathic manipulative treatment (OMT) for patients with low back pain — http://www.guideline.gov/content.aspx?id=15271&search=osteopathic